CLINICAL TRIAL: NCT06225882
Title: Retrospective and Prospective Follow-up of Patients With Primary Hyperoxaluria Type 1 Treated With Lumasiran in France - DAILY-LUMA
Brief Title: Retrospective and Prospective Follow-up of Patients With Primary Hyperoxaluria Type 1 Treated With Lumasiran in France.
Acronym: DAILY-LUMA
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0535
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Patients With PH1 Treated With Lumasiran in France
Keywords: lumarisan; Primary hyperoxaluria type 1 (PH1); retrospective and prospective data.
MeSH Terms: conditions — Primary hyperoxaluria type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lumasiran: Patient with primary hyperoxaluria type 1 who has been treated with Lumasiran, since the beginning of the ATU (temporary authorization for use) and in post-marketing.
  Interventions: Drug: Oxaluria evolution.

INTERVENTIONS:
Drug: Oxaluria evolution. — To collect real data from the specific French experience by collecting data from patients treated throughout the country and to monitor in particular the evolution of oxaluria before and after treatment.

SUMMARY:
Primary hyperoxaluria type 1 (PH1) is a rare genetic disease caused by mutation in the AGXT gene encoding the hepatic peroxisomal enzyme AGT. Reduced AGT activity results in increased glyoxylate and oxalate production, causing the formation of kidney stones, nephrocalcinosis and renal failure. Clinical trials of Lumasiran have provided information on the efficacy and safety of Lumasiran in the treatment of primary hyperoxaluria type 1. However, they do not provide data on long-term efficacy, safety and patient management. As part of the post-marketing follow-up of Lumasiran, in agreement with the authorities, this study proposes a retrospective and prospective follow-up over 5 years of pediatrics and adults patients treated in France with a standardized clinical, biological and radiological follow-up. The main objective is to monitor the evolution of PH1 parameters and particularly oxaluria before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient with primary hyperoxaluria type 1 who has been treated with Lumasiran, since the beginning of the ATU (temporary authorization for use) and in post-marketing.

Exclusion Criteria:

* Opposition of the patient or his legal representatives for minors.
* Not covered by social security.

Ages: 0 Years to 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patient with primary hyperoxaluria type 1 who has been treated with Lumasiran in France.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evolution of oxaluria. | At baseline, At 1 month from the baseline, At 2 months from baseline, At 3 months from baseline, At 6 months from baseline, At 9 months from baseline, At 12 months from baseline, At 18 months from baseline, And 2 times a year until 5 year
  The evolution of oxaluria is followed by urinary biological analysis.

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CHU de Besançon, Besançon
  - Centre de Référence des Maladies Rénales Rares - Hospices Civils de Lyon - Service de Néphrologie et Rhumatologie Pédiatriques - Hôpital Femme Mère Enfant, Bron
  - Hopital Edouard Herriot, Lyon
  - AP-HM - Timone Enfants, Marseille
  - Hôpital Européen G. Pompidou, Paris
  - CHU Paris - Hôpital Necker-Enfants Malades, Paris
  - Hôpital Necker, APHP Paris, Service de néphrologie-dialyse, 149 rue de Sèvres, Paris, Île-de-France Region